CLINICAL TRIAL: NCT01477944
Title: Pattern of Statins Use in Catalonia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CES-CRE-2011/1
Record Dates: First submitted 2011-11-18; First posted 2011-11-23 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Hypercholesteremia
Keywords: Statins pattern of use; Hypercholesterolemic patients; Statins
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To describe the new statins prescription pattern in Catalonia (getting their first prescription for any statin, or receiving a change in their statin treatment including switching, changing in doses or adding ezetimibe/fibrates) since September 2009.

DETAILED DESCRIPTION:
Pattern of statins use in Catalonia.

ELIGIBILITY:
Inclusion Criteria

* Patient with a new prescription of statin Patients receiving one or more changes of the statins treatment

Exclusion Criteria

* Patient with not full information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypercolesterolemic patients in treatment with statins.
Sampling Method: Non-Probability Sample
Enrollment: 180723 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Description of detailed clinical treatment in terms of duration of treatment, doses, drug switches and add-on therapy, in patients with hypercholesterolemia and on treatment with statins from the index date. | From 1st September 2009 to 30th August 2010
Type of prescriber | From 1st September 2009 to 30th August 2010
  Number of patient, whom the drug was prescribed by the specified type of prescriber (specialist, general practitioner, etc.)
Date of change from previous statin to new. | From 1st September 2009 to 30th August 2010

SECONDARY OUTCOMES:
Description of demographic data including: Sex, Age, Height (cm), Weight (kg), Smoking habits (packs-years), Alcohol consume habits (units/week), active worker or retired, Pregnancy. | From 1st September 2009 to 30th August 2010
Total cholesterol | From 1st September 2009 to 30th August 2010
  Total Cholesterol data was collected till the last laboratory values before the date of change from previous statin to new statin.
  That values will be collected for all the patients fulfilling criteria.
Low Density Lipoprotein (LDL) cholesterol concentration | From 1st September 2009 to 30th August 2010
  LDL cholesterol data was collected till the last laboratory values before the date of change from previous statin to new statin.
High Density Lipoproteins (HDL) cholesterol concentration | From 1st September 2009 to 30th August 2010
  HDL data was collected till the last laboratory values before the date of change from previous statin to new statin.
Triglicerides (TG) concentration | From 1st September 2009 to 30th August 2010
  TG data was collected till the last laboratory values before the date of change from previous statin to new statin.
Aspartate Aminotransferase (ASAT) concentration | From 1st September 2009 to 30th August 2010
  ASAT data was collected till the last laboratory values before the date of change from previous statin to new statin.
Serum Glucose concentration | From 1st September 2009 to 30th August 2010
  Serum Glucose data was collected till the last laboratory values before the date of change from previous statin to new statin.
Serum Creatin Kinase (CK) concentration | From 1st September 2009 to 30th August 2010
  CK data was collected till the last laboratory values before the date of change from previous statin to new statin.